CLINICAL TRIAL: NCT03119753
Title: Dimensional Accuracy of Maxillary Complete Denture Base Fabricated by Rapid Prototyping Method Compared With the Conventional Method: A Randomized Controlled Trial
Brief Title: Dimensional Accuracy of Complete Denture With Rapid Prototyping and Conventional Method
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Tarek Salah Hashim Ali, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 8790
Record Dates: First submitted 2017-04-11; First posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Stability
Keywords: Rapid Prototyping technique; complete denture

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group R (Experimental): Rapid Prototyping method of fabrication of complete denture: the master casts will be scanned using DENTAL WINGS eco-scan 3, using laser technology for scanning, after spraying the stainless steel pins with scanning spray to be recorded into the denture base. Virtual model will be obtained for fabrication of denture bases. Denture base will be designed and modified on the virtual model, then it will be printed using ZENITH-3D Printer using Urethane acrylate oligomer based photo-polymerized resin.
  Interventions: Device: Rapid Prototyping method of fabrication of complete denture
- Group C (Active Comparator): Conventional method of fabrication of complete denture: Self-cured acrylic resin trial denture bases will be constructed on the obtained master casts, then processing of the final denture bases by conventional clamping method cured by long curing cycle (74º C for 8 hours) using heat-cured poly-methyl methacrylate (PMMA) resin material. The position of the pins will be recorded into the denture bases so that the linear changes could be measured.
  Interventions: Device: Conventional method of fabrication of complete denture

INTERVENTIONS:
Device: Rapid Prototyping method of fabrication of complete denture — For Rapid Prototyping Method of fabrication of complete denture : the master casts will be scanned using DENTAL WINGS eco-scan 3, using laser technology for scanning, after spraying the stainless steel pins with scanning spray to be recorded into the denture base. Virtual model will be obtained for fabrication of denture bases. Denture base will be designed and modified on the virtual model, then it will be printed using ZENITH-3D Printer using Urethane acrylate oligomer based photo-polymerized resin.
  Arms: Group R
Device: Conventional method of fabrication of complete denture — For Conventional Method of fabrication of complete denture: Self-cured acrylic resin trial denture bases will be constructed on the obtained master casts, then processing of the final denture bases by conventional clamping method cured by long curing cycle (74º C for 8 hours) using heat-cured poly-methyl methacrylate (PMMA) resin material. The position of the pins will be recorded into the denture bases so that the linear changes could be measured.
  Arms: Group C

SUMMARY:
In this study we are going to compare dimensional accuracy of maxillary complete denture base fabricated by using rapid prototyping method and conventional method.

We hypothesize that both techniques do not significantly differ from each other

DETAILED DESCRIPTION:
The study will be carried out in the department of prosthodontics, Faculty of Oral and Dental Medicine, Cairo University. Fourteen patients will be selected from the out-patient clinic according to the inclusion and exclusion criteria, the participants will be divided randomly into two equal groups. The clinical procedures on denture fabrication for both groups will be carried out by TS. The laboratory steps will be carried out by one well trained dental technician (MA). The set of dentures will be fabricated according to the conventional method (Group C) as follow: First appointment: preliminary impression will be obtained by using irreversible hydrocolloid (alginate, cavex, normal set) in stainless steel stock trays. Trays will be augmented with warm utility wax strips (cavex) and shaped by tongue movements and manipulation of labial and buccal tissues. A special tray will be prepared with self-cured acrylic resin (Acrostone-Egypt) over the study cast poured from preliminary impression. Second appointment: A secondary impression will be made with putty rubber base as a border molding material and the final impression will be made with medium rubber base impression material. The final impressions will be poured with type 4 Hydrocal dental stone (Hydrocal Dental stone, Moldano, Bayer Leverkusen, and Germany) to obtain the master cast which will be used for constructing self-cured acrylic resin trial denture bases that will carry a wax occlusion rim. Third appointment: A face bow record will be made to transfer the relation of the maxilla to the temporomandibular joint. Maxilla-mandibular relationship will be recorded using maxillary and mandibular occlusion rims formed over the master cast. Fourth appointment: Setting of artificial teeth will be performed and trial dentures will be tried in inside patients' mouth. Fifth appointment: The finished and polished dentures will be delivered immediately after the necessary adjustments and instructions regarding hygiene and maintenance. The other set of dentures (Group R) will be fabricated according to the rapid prototyping Stereo lithography (SLA) method. The detailed procedures are the same as described for the conventional method (Group C) except for that master casts will be scanned to fabricate the denture bases. The obtained master casts will be used to attach three stainless steel pins before fabrication of the denture bases to assess the linear dimensional changes at the following positions; A: pin at the incisive papilla B: pin at the right second molar area C: pin at the left second molar area Digital caliper will be used to measure distance between the points (AB, BC and CA) and each measurement will be repeated five times. The mean of five readings will be taken as a single reading to decrease the percentage of error. For Conventional Methods: Self-cured acrylic resin trial denture bases will be constructed on the obtained master casts, then processing of the final denture bases by conventional clamping method cured by long curing cycle (74º C for 8 hours) using heat-cured poly-methyl methacrylate (PMMA) resin material. The position of the pins will be recorded into the denture bases so that the linear changes could be measured. For Rapid Prototyping Method: the master casts will be scanned using DENTAL WINGS eco-scan 3, using laser technology for scanning, after spraying the stainless steel pins with scanning spray to be recorded into the denture base. Virtual model will be obtained for fabrication of denture bases. Denture base will be designed and modified on the virtual model, then it will be printed using ZENITH-3D Printer using Urethane acrylate oligomer based photo-polymerized resin. After finishing and polishing of the conventional denture bases and printing of rapid prototyped denture bases, evaluation of linear dimensional changes will be carried out through recording five reading for each of the three dimensions and a mean value will be calculated using digital caliper. This value will be calculated for the master model. The same procedure will be repeated for the two experimental groups (A&B). The dimensional changes will be determined based on the difference between the two values for each method and all records will be tabulated and analysis will be done for the differences between records.

ELIGIBILITY:
Inclusion Criteria:

* Age ranging from 40-70 years.
* Class I Angle's ridge relationship.
* Literate patients are able to understand and respond to a written questionnaire in Arabic.
* Cooperative patients with no history psychological diseases.
* A period of at least six months should elapse from the last extraction.

Exclusion Criteria:

* Pathological changes of residual ridges.
* Patients with debilitating systemic diseases.
* Patients with xerostomia.
* Patients with temporo-mandibular joint disorders or systemic or neuromuscular disorder that might affect chewing efficiency of masticatory muscles.
* Patients with macroglossia or microstomia
* Patients with flabby and flat ridges.
* Patients with allergy to acrylic resin

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2017-06-10 (Estimated); Primary Completion 2017-07-10 (Estimated); Study Completion 2017-09-10 (Estimated)

PRIMARY OUTCOMES:
dimensional accuracy of complete denture | 1 month
  dimensional accuracy of complete denture will be measured using digital caliper

IPD SHARING:
Plan to Share IPD: Undecided